CLINICAL TRIAL: NCT00003022
Title: Phase I Study of Intrathecal 131-I-3F8 Monoclonal Antibody in Patients With GD2 Positive Leptomeningeal Neoplasms
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Leptomeningeal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-021; CDR0000065607 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1267
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Brain and Central Nervous System Tumors; Intraocular Melanoma; Lung Cancer; Melanoma (Skin); Neuroblastoma; Retinoblastoma; Sarcoma
Keywords: metastatic osteosarcoma; childhood infratentorial ependymoma; recurrent childhood rhabdomyosarcoma; childhood supratentorial ependymoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; recurrent neuroblastoma; retinoblastoma; intraocular retinoblastoma; extraocular retinoblastoma; recurrent retinoblastoma; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent osteosarcoma; recurrent adult brain tumor; iris melanoma; ciliary body and choroid melanoma, small size; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; recurrent intraocular melanoma; adult brain stem glioma; adult medulloblastoma; stage IV melanoma; recurrent melanoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; localized unresectable neuroblastoma; adult ependymoblastoma; recurrent childhood brain stem glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood visual pathway glioma; recurrent childhood medulloblastoma; recurrent childhood visual pathway and hypothalamic glioma; previously treated childhood rhabdomyosarcoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood ependymoma; adult oligodendroglioma; adult anaplastic astrocytoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult diffuse astrocytoma; adult pilocytic astrocytoma; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Uveal Melanoma; Lung Neoplasms; Melanoma; Neuroblastoma; Retinoblastoma; Sarcoma; Osteosarcoma; Small Cell Lung Carcinoma; Brain Neoplasms; Medulloblastoma; Ependymoma; Oligodendroglioma; Glioma; Neuroectodermal Tumors, Primitive; Optic Nerve Glioma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma; Astrocytoma; Glioblastoma; Gliosarcoma

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody 3F8

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have leptomeningeal metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the clinical toxicities of intrathecal iodine I 131 monoclonal antibody 3F8 (I-3F8) in patients with GD2 positive leptomeningeal neoplasms.
* Determine whether I-3F8 can detect GD2 positive leptomeningeal tumors.
* Measure the cerebrospinal fluid (CSF) levels and serum pharmacokinetics of I-3F8 in these patients.

OUTLINE: This is a dose escalation study.

Patients receive a single injection of intraventricular or intrathecal iodine I 131 monoclonal antibody 3F8. Patients without objective disease progression and no grade 3 or 4 toxicity 6 weeks after the first dose may receive a second injection.

Cohorts of at least 3 patients are entered at escalating doses of I-3F8. If grade 3 or worse toxicity occurs in 1 or more of 3 patients at a given dose level, then 3 additional patients are accrued at that level. If 2 or more of 6 patients at a given dose level experience grade 3 or worse toxicity, then that dose is declared the maximum tolerated dose (MTD).

Patients are followed weekly for 4 weeks.

PROJECTED ACCRUAL: Approximately 3-30 patients will be accrued for this study over 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy expressing GD2, including, but not limited to:

  * Medulloblastoma/primitive neuroectodermal tumor of the CNS
  * Malignant glioma
  * Neuroblastoma
  * Retinoblastoma
  * Ependymoma
  * Sarcoma
  * Melanoma
  * Small cell lung carcinoma
  * Other tumor types must have GD2 expression confirmed by immunohistochemical staining
* Cerebrospinal fluid or leptomeningeal disease that is refractory to conventional therapy or for which no conventional therapy exists
* Prior measurable human anti-mouse monoclonal antibody titer allowed

PATIENT CHARACTERISTICS:

Age:

* 3 and over

Performance status:

* Not specified

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin less than 3 mg/dL

Renal:

* Creatinine less than 2 mg/dL
* Blood urea nitrogen less than 30 mg/dL

Other:

* May have active malignancy outside the central nervous system
* No obstructive hydrocephalus
* No CNS grade 3 or 4 toxicity as a consequence of prior treatments
* No life threatening infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior monoclonal antibody treatment allowed

Chemotherapy:

* Prior chemotherapy allowed
* Must have recovered from all hematopoietic and neurologic side effects of prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed
* At least 6 weeks since prior cranial or spinal irradiation

Surgery:

* Not specified

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-04; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Kramer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Kramer K, Humm JL, Souweidane MM, Zanzonico PB, Dunkel IJ, Gerald WL, Khakoo Y, Yeh SD, Yeung HW, Finn RD, Wolden SL, Larson SM, Cheung NK. Phase I study of targeted radioimmunotherapy for leptomeningeal cancers using intra-Ommaya 131-I-3F8. J Clin Oncol. 2007 Dec 1;25(34):5465-70. doi: 10.1200/JCO.2007.11.1807. PMID 18048828